CLINICAL TRIAL: NCT00741819
Title: An Open Label, Multi-center Study Evaluating the Safety of Long-term Inhaled Treprostinil Administration Following Transition From Inhaled Ventavis® (Iloprost) in Subjects With Pulmonary Arterial Hypertension.
Brief Title: Safety Evaluation of Inhaled Treprostinil Administration Following Transition From Inhaled Ventavis in Pulmonary Arterial Hypertension (PAH) Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIN-PH-401
Record Dates: First submitted 2008-08-23; First posted 2008-08-26 (Estimated); Results first posted 2013-02-20 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; PAH; treprostinil sodium; inhalation; ventavis; iloprost
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Respiratory Aspiration | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inhaled treprostinil (Experimental): Solution for oral inhalation treprostinil (0.6 mg/mL). Inhaled via an ultrasonic nebulizer which provides a dose of 6mcg of treprostinil per breath. Doses are titrated up to 12 breaths four times daily.
  Interventions: Drug: Inhaled treprostinil

INTERVENTIONS:
Drug: Inhaled treprostinil
  Other Names: Tyvaso

SUMMARY:
This is a 24-month, multi-center, prospective, open-label, safety evaluation in PAH subjects following transition from a stable dose of inhaled iloprost (Ventavis).

Subjects are to be evaluated for safety throughout the course of the study while secondary assessments will be conducted at Baseline, Week 6, Week 12, and Months 6, 12, 18 and 24 following initiation of treprostinil sodium.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 75 years of age
* PAH diagnosis defined by following WHO Group I categories: idiopathic/familial, associated with unrepaired or repaired congenital systemic-to-pulmonary shunts (repaired >/= 5 years), associated with collagen vascular disease, associated with HIV, associated with appetite suppressant/toxin use
* Baseline six-minute walk distance (6MWD) >/= 250 meters
* Currently receiving Ventavis and be stable at current dose for 30 days prior to Baseline
* If currently receiving other approved background therapy (i.e. endothelin receptor antagonist or phosphodiesterase-5-inhibitor or both) must be on stable dose for 30 days prior to Baseline
* Previous testing (e.g. right heart catheterization, echocardiography) consistent with diagnosis of PAH

Exclusion Criteria:

* Nursing or pregnant
* Has acute concomitant disease (e.g. portal hypertension, chronic thromboembolic disease, pulmonary veno-occlusive disease, etc) other than those accepted as part of the inclusion criteria or has had atrial septostomy
* History of uncontrolled sleep apnea, left-sided heart disease, or parenchymal lung disease
* Use of investigational drug within 30 days of Baseline

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-09; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - University of Alabama Birmingham, Birmingham, Alabama
  - UCSD Medical Center, La Jolla, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Kansas University Medical Center, Kansas City, Kansas
  - Long Island Jewish Medical Center - North Shore, New Hyde Park, New York
  - Beth Israel Medical Center, New York, New York
  - Cornell University Medical Center, New York, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - Mary M. Parkes Center for Asthma, Allergy and Pulmonary Care, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began 09-Dec-2008 and ended 09-Mar-2010. All recruitment took place in medical clinic settings.
Pre-assignment Details: Not applicable given this was an open-label study.
Groups:
- Inhaled Treprostinil: Inhaled treprostinil was given four times daily at doses titrated up to 12 breaths.
Period: Overall Study
Arm/Group | Inhaled Treprostinil
Started | 73
Completed | 65
Not Completed | 8
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 3
Not completed — Death | 1
Not completed — Disease progression | 1

BASELINE CHARACTERISTICS:
Groups:
- Inhaled Treprostinil: Inhaled treprostinil was titrated up to 12 breaths four times daily.
Arm/Group | Inhaled Treprostinil
Number analyzed (Participants) | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 63
  >=65 years | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 49.4 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 73
Pulmonary Arterial Hypertension (PAH) etiology [Number; unit: participants]
  Idiopathic PAH or familial PAH | 35
  Connective Tissue Diseases (CTD) | 16
  Congenital heart disease (CHD)-repaired shunt | 4
  CHD-unrepaired shunt | 15
  HIV | 3
Background PAH therapy [Number; unit: participants]
  None | 3
  Endothelin receptor antagonist (ERA) | 19
  Phosphodiesterase-5 inhibitor (PDE-5i) | 8
  ERA and PDE-5i | 43
Six-minute walk distance (6MWD) [Median (Full Range); unit: meters] | 378 (78) [259 to 600]
N-terminal prohormone brain natriuretic peptide (NT-proBNP) [Median (Full Range); unit: pg/mL] | 626 [26 to 8324]

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Overall safety of transitioning from inhaled iloprost to inhaled treprostinil was assessed by type and frequency of adverse events.
Time Frame: up to 24 months
Population: All subjects who received at least one dose of inhaled treprostinil were included in the safety analysis population.
Measure: Number; unit: number of events
Groups:
- Inhaled Treprostinil: up to 12 breaths four times daily
Arm/Group | Inhaled Treprostinil
Number analyzed (Participants) | 73
number of events
  Overall events | 440
  Possibly or Probably related events | 266
  Severe events | 41
  Serious events | 15

2. Secondary Outcome: Six-minute Walk Distance (6MWD)
Description: Change in 6MWD from Baseline to Week 12. The 6-minute walk test (6MWT) was conducted at Baseline (10-30 minutes following the last dose of inhaled iloprost) and at Week 12 (10-60 minutes following the dose of inhaled treprostinil). The change in distance (meters) between Baseline and Week 12 is reported below.
Time Frame: Baseline and 12 weeks
Population: Subjects enrolled at Week 12 visit.
Measure: Median (Full Range); unit: meters
Arm/Group | Inhaled Treprostinil
Number analyzed (Participants) | 68
meters
  Week 12 | 392.5 [220 to 708]
  Change from Baseline | 16 (78) [-51 to 108]
Statistical Analysis 1: Comparison: Inhaled Treprostinil; Analysis of endpoints was descriptive in nature. Numeric endpoints for post-baseline assessments were compared to Baseline using Wilcoxon signed rank test, and p-values were calculated for descriptive purposes; no formal hypothesis testing was planned; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank test]; Median Difference (Final Values) = 16, Standard Deviation 35.9 — Change in 6MWD from Baseline was calculated for patients still remaining on study at Week 12

3. Secondary Outcome: Quality of Life (QoL) Assessment: Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR)
Description: Change in CAMPHOR Scores from Baseline to Week 12. The CAMPHOR is a health related quality of life instrument validated for pulmonary hypertension that assesses impairment (symptoms), disability (activities) and quality of life. The questionnaire is divided into three sections; Symptoms (Scores 0-25; high scores indicate more symptoms), Activity (Score 0-30; low score indicates good functioning)and Quality of Life (0-25; high scores indicate poor QoL). The sum of these scores equates to the Total score (0-80). In the CAMPHOR scores, lower scores indicate improvements.
Time Frame: Baseline and 12 weeks
Population: Subjects who were still enrolled and completed the questionnaire at Baseline and Week 12. Total analysis population was less for the activity score and total score (N = 67).
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Inhaled Treprostinil
Number analyzed (Participants) | 69
units on a scale
  Symptom Score at Week 12 | 5.3 [0 to 21]
  Change in Symptom Score | -2.9 (3.9) [-13 to 8]
  Activity Score at Week 12 | 6.6 [0 to 16]
  Change in Activity Score | -1.2 (2.5) [-9 to 5]
  Quality of Life Score at Week 12 | 4.9 [0 to 20]
  Change in Quality of Life Score | -2.4 (3.9) [-14 to 5]
  Total Score at Week 12 | 16.8 [0 to 53]
  Change in Total Score | -6.4 (7.7) [-29 to 7]
Statistical Analysis 1: Comparison: Inhaled Treprostinil; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank test; Mean Difference (Final Values) = -6.4, Standard Deviation 7.7 — Analysis based on Total CAMPHOR Score

4. Secondary Outcome: Treatment Satisfaction Questionnaire of Medication (TSQM)
Description: Change in TSQM score from Baseline to Week 12. The TSQM is a validated instrument (Health and Quality of Life Outcomes 2004, 2:12) that measures major dimensions of patient satisfaction with medications. The questionnaire is comprised of 15 questions which fall into one of four categories; Effectiveness, Side-Effects, Convenience, and Global Satisfaction. Responses are scaled on a seven point bipolar scale from 'Extremely Satisfied' to 'Extremely Dissatisfied' where higher scores indicate improvements (total scores from 0-100). The questionnaire was completed at Baseline and Week 12. The Baseline questionnaire focused on the subject's satisfaction with inhaled iloprost treatment, while the questionnaire completed at Week 12 focused on the subject's satisfaction with inhaled treprostinil.
Time Frame: Baseline and 12 weeks
Population: Subjects who completed the TSQM at Baseline and Week 12. Total analysis population was less for the Convenience Score (N=67) and Global Satisfaction Score (N=66).
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Inhaled Treprostinil
Number analyzed (Participants) | 68
units on a scale
  Effectiveness Score at Week 12 | 81.9 [44 to 100]
  Change in Effectiveness Score | 19.9 (21.5) [-28 to 94]
  Side-effects Score at Week 12 | 84.4 [25 to 100]
  Change in Side-Effects Score | -0.5 (21.3) [-75 to 56]
  Convenience Score at Week 12 | 83.3 [33 to 100]
  Change in Convenience Score | 38.3 (25.9) [0 to 100]
  Global Satisfaction Score at Week 12 | 81.9 [36 to 100]
  Change in Global Satisfaction | 20.0 (23.7) [-36 to 100]
Statistical Analysis 1: Comparison: Inhaled Treprostinil; Test type: Superiority or Other; p = 0.895, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.5, Standard Deviation 21.3 — Side-Effects Score, change from Baseline to Week 12
Statistical Analysis 2: Comparison: Inhaled Treprostinil; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test; Mean Difference (Final Values) = 38.3, Standard Deviation 25.9 — Convenience Score, change from Baseline to Week 12
Statistical Analysis 3: Comparison: Inhaled Treprostinil; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test; Mean Difference (Final Values) = 20.0, Standard Deviation 23.7 — Global Satisfaction, change from Baseline to Week 12
Statistical Analysis 4: Comparison: Inhaled Treprostinil; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank test; Mean Difference (Final Values) = 19.9, Standard Deviation 21.5 — Effectiveness score, change from Baseline to Week 12

5. Secondary Outcome: Patient Impression of Change
Description: The patient impression of change (PIC) was three single therapy-related questions related to the subjects overall impression of the transition from inhaled iloprost to inhaled treprostinil. Subjects were surveyed related to their overall impression of the transition from inhaled iloprost to inhaled treprostinil at Week 12.
Time Frame: Baseline and 12 weeks
Population: Subjects who completed questionnaire at Baseline and Week 12
Measure: Number; unit: percentage of patients
Arm/Group | Inhaled Treprostinil
Number analyzed (Participants) | 67
percentage of patients
  Improvement of Symptoms | 73 (80.5)
  Improvment in Time Spent | 91
  Overall Satisfaction | 94

6. Secondary Outcome: N-terminal Prohormone of Brain Natriuretic Peptide (NT-proBNP)
Description: Change in NTpro-BNP from Baseline to Week 12. Blood samples were collected for plasma NTpro-BNP analysis during the study.
Time Frame: Baseline and Week 12
Population: Subjects with a NTproBNP sample drawn at Baseline and Week 12
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Inhaled Treprostinil
Number analyzed (Participants) | 68
pg/mL | -74 [-4728 to 3837]
Statistical Analysis 1: Comparison: Inhaled Treprostinil; Test type: Superiority or Other; p = 0.001, Wilcoxon signed-rank test

7. Secondary Outcome: World Health Organization (WHO) Functional Class
Description: Change in WHO Functional Class (FC) from Baseline to Week 12. Data presented as percent of subjects who either improved FC, worsened FC, or had no change in FC from Baseline to Week 12.
Time Frame: Baseline and 12 Weeks
Population: Subjects still enrolled at Week 12 with a WHO Functional Class at Baseline and Week 12.
Measure: Number; unit: percentage of subjects
Arm/Group | Inhaled Treprostinil
Number analyzed (Participants) | 69
percentage of subjects
  Improvement | 6
  No Change | 87
  Worsened | 7

8. Secondary Outcome: Drug Administration Activities Questionnaire
Description: Change in tasks from Baseline to Week 12. At Baseline and Week 12, subjects provided information related to the daily administration and time requirements of inhaled iloprost (Baseline) and inhaled treprostinil (Week 12).
Time Frame: Baseline and 12 weeks
Population: Subjects who completed the questionnaire at Baseline and Week 12.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Inhaled Treprostinil
Number analyzed (Participants) | 61
minutes
  Week 12 Total Daily Dosing Time | 39.1 (25.1)
  Change in Time Total Daily Dosing Time | -79.3 (80.5)

ADVERSE EVENTS:
Time Frame: up to 56 weeks
Arm/Group | Inhaled Treprostinil
Serious Adverse Events (participants affected / at risk) | 10/73
Other Adverse Events (participants affected / at risk) | 71/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Treprostinil (N=73)
Pneumonia (Infections and infestations) | 2 (2)
Pulmonary hypertension (Cardiac disorders) | 2 (2)
Cor pulmonale (Cardiac disorders) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
psychotic disorder (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Treprostinil (N=73)
Cough (Respiratory, thoracic and mediastinal disorders) | 54 (55)
Headache (Nervous system disorders) | 32 (32)
Nausea (Gastrointestinal disorders) | 22 (23)
Chest discomfort (General disorders) | 12 (12)
upper respiratory tract infection (Infections and infestations) | 11 (13)
nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 11 (12)
flushing (Vascular disorders) | 11 (11)
dizziness (Nervous system disorders) | 10 (13)
palpitations (Cardiac disorders) | 9 (9)
throat irritation (Respiratory, thoracic and mediastinal disorders) | 9 (9)
fatigue (General disorders) | 8 (8)
productive cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7)
diarrhea (Gastrointestinal disorders) | 6 (6)
bronchitis (Infections and infestations) | 5 (5)
chest pain (General disorders) | 5 (5)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
pain in jaw (Musculoskeletal and connective tissue disorders) | 5 (5)
rash (Skin and subcutaneous tissue disorders) | 5 (5)
somnolence (Nervous system disorders) | 5 (5)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
fluid retention (Metabolism and nutrition disorders) | 4 (4)
pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
sinusitis (Infections and infestations) | 4 (4)

LIMITATIONS AND CAVEATS:
Small, open-label study without comparison arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the United Therapeutics publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.